CLINICAL TRIAL: NCT06833424
Title: Predictors of Dural Venous Sinus Stenting in Idiopathic Intracranial Hypertension Patients and Outcomes
Brief Title: Dural Venous Sinus Stent in Idiopathic Intracranial Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Zayed Saber, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: intracranial hypertension
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: predictors and outcomes
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dural Venous sinus stent (Experimental): 40 Patients Diagnosed with idiopathic intracranial hypertension according to modified Dandy Criteria subjected to Dural venous sinus stenting
  Interventions: Procedure: Dural venous sinus stenting

INTERVENTIONS:
Procedure: Dural venous sinus stenting — 40 patients with idiopathic intracranial hypertension according to Modified Dandy Criteria will subjected to Dural venous stenting

SUMMARY:
This study aims to identify clinical determinants and factors that predict outcome including primary outcome and secondary outcome depending on factors in individual patients with Idiopathic intracranial hypertension treated by Dural venous sinus stenting.

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) has long been associated with the hallmark clinical triad of headaches, papilledema, and visual loss in the absence of neurologic signs (except possible CN VI palsy), Hydrocephalus or intracranial masses on CT or MRI. findings without evidence of thrombosis; lumbar puncture opening pressure of >25 cmH2O; normal biochemical and cytological composition of the CSF. The overall age-adjusted and gender-adjusted annual incidence is increasing and was reported to be 2.4 per 100 000 within the last decade (2002-2014).A variety of aetiologies have been suggested to explain the pathophysiology behind IIH, including meningeal inflammation, metabolic disturbances (e.g., hyper- or hypoadrenalism and hypoparathyroidism), medication effects (e.g., excess vitamin A, corticosteroids, and tetracycline), and cerebral venous hypertension.Imaging of patients with IIH is traditionally performed to exclude lesions that produce intracranial hypertension. MR imaging features of IIH include posterior globe flattening, a protrusion of the subarachnoid space in the cavum sellae (Empty Sella), distension of the preoptic subarachnoid space, enhancement of the prelaminar optic nerve, vertical tortuosity of the orbital optic nerve, and intraocular protrusion of the prelaminar optic nerve. Although these findings support the presence of elevated ICP and, thus, the diagnosis of IIH, they are not predictive of the severity of visual loss, and their absence does not exclude the diagnosis. It should not guide a specific management of patients with IIH .

The first line of treatment for IIH consists of weight loss and/or medical therapy including diuretics such as acetazolamide. When medical treatment fails, surgical options include cerebrospinal fluid (CSF) diversion via ventriculoperitoneal (VP) or lumboperitoneal (LP) shunting or optic nerve sheath fenestration. Recently, another etiology of cerebral venous hypertension has garnered increasing attention as a putative cause of IIH, cerebral venous Dural sinus stenosis. In medically refractory IIH patients with a physiologic pressure gradient across venous stenosis, cerebral venous stenting has emerged as an alternative treatment to traditional surgical approaches.

Transverse sinus stenosis can be seen in 2 morphologic forms: an extrinsic smooth gradually narrowing tapered stenosis and intrinsic discrete obstructions, presumably due to arachnoid granulations or fibrous septae. While intrinsic transverse sinus stenosis might cause IIH by completely occluding the transverse sinus, the extrinsic compression resolves with CSF drainage. might be secondary to intracranial hypertension. Venous sinus stenting (VSS) reduces intracranial venous pressures and improves idiopathic intracranial hypertension (IIH) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 40 Patients of idiopathic intracranial hypertension subjected to Dural venous sinus stenting met the modified Dandy criteria for (IIH).

  1. Signs and symptoms of increased intracranial pressure: Headaches, nausea, vomiting, visual changes, and papilledema.
  2. No localizing or focal neurologic signs: Except for possible unilateral or bilateral VI nerve paresis.
  3. Elevated cerebrospinal fluid (CSF) pressure: Without cytologic or chemical abnormalities.
  4. No etiology for increased intracranial pressure: On neuroimaging findings.

     * Age: 18-60 years
     * Gender: Male or Female Inclusion Criteria.

Exclusion Criteria

1. Age less than or equal to 18 years.
2. severe allergic reaction to iodine contrast or chronic Kidney disease.
3. contraindication to general anesthesia or antiplatelet anticoagulants, Hemorrhagic Diathesis
4. patients with secondary causes of intracranial hypertension: Dural arteriovenous fistula or other arteriovenous lesion affecting cortical venous flow.
5. pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
change in headache impact scale(HIT-6) | 3, 6 months
  The Headache Impact Test (HIT) is a tool used to measure the impact headaches have on your ability to function on the job, at school, at home and in social situations. Your score shows you the effect that headaches have on normal daily life and your ability to function. minimum score 36 and maximum score 78
Papilledema Friesen grading scale | 3 months and 6 months
  The Frisen grading system is an objective criteria used to describe the degree of papilledema, which is swelling of the optic disc from increased ICP grading from zero to 5
Visual filed Assessment Perimetry | 3,6 months
  Perimetry is the systematic measurement of visual field function (the total area where objects can be seen in the peripheral vision while the eye is focused on a central point).
Changes in other symptoms tinnitus, abducent nerve palsy and Transient visual Obsecuration | 3,6 months
  changes in other symptomology including tinnitus ,abducent nerve palsyand TVO

SECONDARY OUTCOMES:
Stent Patency and pressure change | 6 months
  Diagnostic DSA follow up and measuring pressure gradient changes pre and post stenting
stent Patency | 6 months
  in stent stenosis and Adjacent stent stenosis
Safety outcome measures | 10 days
  Safety outcomes of occurrences of complication: Subdural Hematoma, Subarachnoid Hemorrhage, Intracerebral hematoma puncture site complication (retroperitoneal hematoma or femoral artery aneurysm)
Quality of life improvement | 3,6 months
  Quality of life measure: SF-36 for fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Result] Hilvert AM, Gauhar F, Longo M, Grimaudo H, Dugan J, Mummareddy N, Chitale R, Froehler MT, Fusco MR. Venous sinus stenting versus ventriculoperitoneal shunting: comparing clinical outcomes for idiopathic intracranial hypertension. J Neurointerv Surg. 2024 Nov 22;16(12):1264-1267. doi: 10.1136/jnis-2024-022174. PMID 39209429
- [Result] McGonigal A, Bone I, Teasdale E. Resolution of transverse sinus stenosis in idiopathic intracranial hypertension after L-P shunt. Neurology. 2004 Feb 10;62(3):514-5. doi: 10.1212/wnl.62.3.514. No abstract available. PMID 14872049
- [Result] Subramaniam RM, Tress BM, King JO, Eizenberg N, Mitchell PJ. Transverse sinus septum: a new aetiology of idiopathic intracranial hypertension? Australas Radiol. 2004 Jun;48(2):114-6. doi: 10.1111/j.1440-1673.2004.01269.x. PMID 15230741
- [Result] Aguilar-Perez M, Martinez-Moreno R, Kurre W, Wendl C, Bazner H, Ganslandt O, Unsold R, Henkes H. Endovascular treatment of idiopathic intracranial hypertension: retrospective analysis of immediate and long-term results in 51 patients. Neuroradiology. 2017 Mar;59(3):277-287. doi: 10.1007/s00234-017-1783-5. Epub 2017 Mar 2. PMID 28255904
- [Result] Saindane AM, Bruce BB, Riggeal BD, Newman NJ, Biousse V. Association of MRI findings and visual outcome in idiopathic intracranial hypertension. AJR Am J Roentgenol. 2013 Aug;201(2):412-8. doi: 10.2214/AJR.12.9638. PMID 23883223
- [Result] Degnan AJ, Levy LM. Pseudotumor cerebri: brief review of clinical syndrome and imaging findings. AJNR Am J Neuroradiol. 2011 Dec;32(11):1986-93. doi: 10.3174/ajnr.A2404. Epub 2011 Jun 16. PMID 21680652
- [Result] Brodsky MC, Vaphiades M. Magnetic resonance imaging in pseudotumor cerebri. Ophthalmology. 1998 Sep;105(9):1686-93. doi: 10.1016/S0161-6420(98)99039-X. PMID 9754178
- [Result] Kilgore KP, Lee MS, Leavitt JA, Mokri B, Hodge DO, Frank RD, Chen JJ. Re-evaluating the Incidence of Idiopathic Intracranial Hypertension in an Era of Increasing Obesity. Ophthalmology. 2017 May;124(5):697-700. doi: 10.1016/j.ophtha.2017.01.006. Epub 2017 Feb 7. PMID 28187976
- [Result] Starke RM, Wang T, Ding D, Durst CR, Crowley RW, Chalouhi N, Hasan DM, Dumont AS, Jabbour P, Liu KC. Endovascular Treatment of Venous Sinus Stenosis in Idiopathic Intracranial Hypertension: Complications, Neurological Outcomes, and Radiographic Results. ScientificWorldJournal. 2015;2015:140408. doi: 10.1155/2015/140408. Epub 2015 Jun 4. PMID 26146651
- [Result] Friedman DI, Jacobson DM. Diagnostic criteria for idiopathic intracranial hypertension. Neurology. 2002 Nov 26;59(10):1492-5. doi: 10.1212/01.wnl.0000029570.69134.1b. PMID 12455560
- [Result] Radhakrishnan K, Ahlskog JE, Garrity JA, Kurland LT. Idiopathic intracranial hypertension. Mayo Clin Proc. 1994 Feb;69(2):169-80. doi: 10.1016/s0025-6196(12)61045-3. PMID 8309269